CLINICAL TRIAL: NCT05737953
Title: Construction of Molecular Diagnostic Marker Models for Pancreatic Cystic Tumors Based on CfDNA Methylation Sequencing and Proteomic Analysis of Pancreatic Cystic Fluid Samples
Brief Title: Construction of Molecular Diagnostic Marker Model for Pancreatic Cystic Tumors Based on Pancreatic Cystic Fluid Samples
Status: Recruiting | Type: Observational
Sponsor: Zhaoshen Li (Other)
Collaborators: Oriental Hepatobiliary Surgery Hospital Affiliated to Naval Military Medical University (Unknown); Zhejiang University (Other); The First Affiliated Hospital of Nanchang University (Other); West China Hospital (Other); LanZhou University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Peking University Cancer Hospital & Institute (Other); First Hospital of China Medical University (Other); First Affiliated Hospital of Guangxi Medical University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); The Second Affiliated Hospital of Baotou Medical College (Other); Shandong Province Third hospital (Other)
Responsible Party: Sponsor-Investigator, Zhaoshen Li, Director of Gastroenterology Department of Changhai Hospital, Changhai Hospital
Organization: Changhai Hospital (Other)
Other Study IDs: WKX2023-02
Record Dates: First submitted 2023-02-05; First posted 2023-02-21 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Neoplasms; DNA Methylation; Proteome
Keywords: Pancreas cystic neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cystic fluid in pancreatic cystic tumour
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Mucinous tumour group
  Interventions: Diagnostic Test: cfDNA methylation sequencing and proteome analysis
- Non-mucinous tumour group
  Interventions: Diagnostic Test: cfDNA methylation sequencing and proteome analysis

INTERVENTIONS:
Diagnostic Test: cfDNA methylation sequencing and proteome analysis — Sequencing of cfDNA methylation and proteomic analysis of two sets of capsular fluid samples

SUMMARY:
The goal of this observational study is to test in patients with cystic tumor of pancreas. The main questions it aims to answer are:

Screening of molecular diagnostic markers for pancreatic cystic tumors by cfDNA methylation sequencing of pancreatic cystic fluid and proteomic assays to distinguish benign from malignant and mucinous/non-mucinous, correlate with pathological features, and find molecular features associated with the degree of malignancy.

Participants will Provide post-operative cyst fluid specimens.

DETAILED DESCRIPTION:
Patients with pancreatic cystic tumors were divided into control, mucinous tumor and non-mucinous tumor groups, and cfDNA molecules and protein molecules that were significantly altered between different groups were found by cfDNA methylation sequencing of pancreatic cystic fluid and proteomic detection techniques. Multi-omics analysis was performed to construct a more efficient molecular diagnostic marker model. Correlating models with pathological features to find molecular features associated with the degree of malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are ≥ 18 years old, regardless of gender;
* Preoperative imaging examination (EUS, CT, MRI) diagnosed cystic mass of pancreas and suspected cystic tumor;
* Subjects voluntarily accepted radical resection of pancreatic cystic tumors;
* Subjects or family members voluntarily sign the informed consent form for clinical research.

Exclusion Criteria:

* The excised sample does not contain cystic components, or the cystic fluid cannot be collected;
* Receive tumor-related treatment (radiotherapy, chemotherapy, immunotherapy, etc.) before operation;
* Receive antibiotic treatment within 1 week before operation;
* Subjects refused to accept radical resection of pancreatic cystic tumor, or had any situation that they could not accept radical resection of pancreatic cystic tumor;
* The subjects or their families refused to sign the informed consent form for clinical research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic cystic tumor
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Types and concentrations of cfDNA and proteins contained in the vesicular fluid | 2023-11-31
  Identification of protein and circulating gene methylation species in cyst fluid and quantification of their concentrations using mass spectrometry. Characterize cfDNA methylation and proteomics of cyst fluid in patients with pancreatic cystic neoplasm (PCN).

SECONDARY OUTCOMES:
Establishment of a diagnostic model for cystic tumors of the pancreas | 2023-11-31
  A machine learning approach was used to further screen for characteristically methylated cfDNA and proteins in PCN patients.Establishment of a diagnostic model for pancreatic cystic tumors.
Establishing a model for the identification of mucus and non-mucus | 2023-11-31
  A machine learning approach was used to further screen for characteristically methylated cfDNA and proteins in PCN patients.To establish a model for the identification of mucinous and non-mucinous.
Development of a progressive benign malignancy prediction model | 2023-11-31
  A machine learning approach was used to further screen for characteristically methylated cfDNA and proteins in PCN patients.Development of a progression benign malignancy prediction model.

CONTACTS AND LOCATIONS:
Overall Officials: Shiyu Li, Principal Investigator — Changhai Hospital; Chengye Pan, Study Chair — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
cfDNA methylation data and proteome analysis data